CLINICAL TRIAL: NCT04902781
Title: A Sequential, Two-Part Study to Evaluate the Clinical Benefit, Safety, Pharmacokinetics, and Pharmacodynamics of AT-007 in Pediatric Patients With Classic Galactosemia (CG)
Brief Title: Clinical Benefit, Safety, PK and PD Study of AT-007 in Pediatric Subjects With Classic Galactosemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Applied Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-007-1002
Record Dates: First submitted 2020-07-14; First posted 2021-05-26 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Classic Galactosemia
Keywords: Galactosemia; Classic Galactosemia
MeSH Terms: conditions — Galactosemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: AT-007 (Experimental): AT-007 The starting dose in Part A will be 5 mg/kg for all age groups. For each age group, Part B of the study will not start until the optimum dose evaluated in Part A has been identified
  Interventions: Drug: AT-007
- Placebo (Placebo Comparator): Placebo given orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AT-007 — Treatment with AT-007 given orally
  Other Names: aldose reductase inhibitor
  Arms: Experimental: AT-007
Other: Placebo — Placebo given orally
  Arms: Placebo

SUMMARY:
This study is designed to assess the clinical benefit as well as the safety, pharmacokinetics (PK), and pharmacodynamics (PD) (reduction of galactitol levels) of AT-007 in pediatric subjects with Classic Galactosemia (CG).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study in pediatric subjects with CG. Children with CG ages 2 through 17 years will be enrolled. The study is designed to assess the clinical benefit using validated, standardized Clinical Outcome Assessments (COAs) as well as the safety, PK, and PD (reduction of galactitol levels) of AT-007 in pediatric subjects with CG. The study consists of 2 main parts, Part A and Part B, and an open-label extension (OLE).

Part A is an intra-patient dose escalation evaluating multiple ascending doses (MAD) of AT-007.

Part B is designed to assess the clinical benefits of long-term administration of AT-007 (at the optimum dose identified in Part A) on validated, standardized COAs.

Open-label extension (OLE) is an active treatment extension for patients who received placebo treatment in Part B.

ELIGIBILITY:
Inclusion:

* Male
* Female non-pregnant
* Female non-lactating subjects aged ≥2 to <18 years.
* Diagnosis of Classic Galactosemia, confirmed by <1% GALT (galactose-1-phosphate uridyltransferase) enzyme activity in erythrocytes, or a historical record of diagnosis of <1% GALT enzyme activity.

Exclusion:

* Male/Female with no significant health problems (other than classic Galactosemia)
* No other disease that would preclude participation in the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Global Statistical Test (GST) | Month 6, Month 12 and Month 18
  The primary endpoint is a GST of four components: 1) Behavioral Symptoms Index of the Behavioral Assessment Scale for Children 3 (BASC-3); 2) Activities of Daily Living from the BASC-3; 3) Oral Expression from the Oral and Written Language Skills-II (OWLS-II); 4) Listening Comprehension from the OWLS-II. Each individual component is also a secondary endpoint on their own with the test and scoring described below in the secondary endpoint section. For the GST, change from baseline using standardized z-scores is calculated for active versus placebo.
Sensitivity Analysis of the Primary Endpoint (GST) with Cognition | Month 6, Month 12 and Month 18
  Sensitivity Analysis adding the National Institutes of Health Toolbox Cognition Battery (NIH-CB) test which measures cognition. NIH-CB is described below in the secondary endpoints. For the GST with cognition, change from baseline using standardized z-scores is calculated for active versus placebo.
Sensitivity Analysis of the Primary Endpoint (GST) with Fine Motor Skills | Month 6, Month 12 and Month 18
  Sensitivity Analysis adding the National Institutes of Health Toolbox Motor Battery (NIH-MB) 9-Hole Pegboard test which measures fine motor skills. NIH-MB is described below in the secondary endpoints. For the GST with fine motor skills, change from baseline using standardized z-scores is calculated for active versus placebo.

SECONDARY OUTCOMES:
Galactitol Level | Month 1, Month 2, Month 3, Month 6, Month 12, and Month 18
  The change from baseline in plasma galactitol (Pharmacodynamic measure)
Behavioral Assessment System for Children-3 [Individual Components] | Month 6, Month 12 and Month 18
  Behavioral Assessment System for Children (BASC-3) has a normal range of 40-60 with the higher score showing more difficulty. There are multiple outcome scores included such as: Behavioral Symptoms Index, Activities of Daily Living, Withdrawal, Adapatability, Adaptive Skills, Socialization, and Functional Impairment Index.
National Institute of Health Toolbox Cognition Battery | Month 6, Month 12 and Month 18
  Change from baseline in the NIH Toolbox Cognition Battery (NIH-CB). The NIH-CB uses multiple tests to evaluate Cognition and consists of tests of multiple constructs to yield individual ranking and demonstrate Cognitive Function Composite, Fluid Cognition Composite Sequence Memory, List Sorting, Pattern Comparison, and Crystallized Cognition Composite, Picture Vocabulary and Reading Recognition. This is standardized normal or 100 with a standard deviation of 10. Higher scores are better.
Archimedes Spiral Drawing Test | Month 6, Month 12 and Month 18
  The Archimedes Spiral Drawing Test evaluates tremor on a scale of 0 (no tremor) to 4 (severe tremor).
National Institute of Health Toolbox Motor Battery | Month 6, Month 12 and Month 18
  NIH Toolbox Motor Battery (NIH-MB) is a multiple of tests to determine fine motor skills using the 9-Hole Pegboard Test and gross motor skills using the Standing Balance Test. This is standardized normal or 100 with a standard deviation of 10. Higher scores are better.
Scale for Assessment & Rating of Ataxia | Month 6, Month 12 and Month 18
  Scale for Assessment & Rating of Ataxia (SARA) is 0-40, the higher the score the worse value
Oral and Written Language Scales-II | Month 6, Month 12 and Month 18
  Oral and Written Language Scales-II (OWLS-II) has both an Oral Expression and Listening Comprehension score. Scores are 0-100 with a standard deviation of 15.
Rate of Lens Opacity | Month 6, Month 12 and Month 18
  Onset and severity/progression of cataracts using the Lens Opacity System (LOCS) III, has a grading scale of 1-4, with 4 the most severe as assessed by the reviewer per standard criteria for anterior and posterior obstruction of the eye.
Sexual maturation in female patients as indicated by Tanner Stage | Month 6, Month 12 and Month 18
  Sexual maturation in female patients as indicated by Tanner Stage 1- 4 which is the ranking of physical development in children, adolescents and adults. This defines physical measurements of development based on external primary and secondary sex characteristics, such as the size of the breasts, and development of pubic hair. This is assessed by physical exam with Stage 1 per-pubescent and Stage 4 post pubescent.
Ovarian function in female patients determined by hormonal tests. | Month 6, Month 12 and Month 18
  Ovarian function in female patients is recorded by hormonal measures: FSH (follicle stimulating hormone), estradiol, and LH (luteinizing hormone).

OTHER OUTCOMES:
Biomarker Analysis [Exploratory] | Month 1, Month 2, Month 3, Month 6, Month 12, and Month 18
  This biomarker analysis will be performed to assess the levels of galactose and its other metabolites; Exploratory Endpoint
Bayley Scales of Infant and Toddler Development-4 [Exploratory] | Month 6, Month 12 and Month 18
  Bayley Scales of Infant and Toddler Development (Bayley-4) showing a score of 40 -160 with higher values showing more development. Exploratory Endpoint
Vineland Adaptive Behavior Scales-3 [Exploratory] | Month 6, Month 12 and Month 18
  Vineland Adaptive Behavior Scales (Vineland-3) has a normal score of 100 and lower scores show developmental delay; Exploratory Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Waisbren, PhD, Study Chair — Harvard University; Jonathan W Mink, MD, Study Chair — University of Rochester
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research Center, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No